CLINICAL TRIAL: NCT07279363
Title: Cognitive Behavioral Therapy for Treatment-Seeking to Improve Treatment Engagement and Reduce Suicide Risk Among Deaf Individuals
Brief Title: Deaf CBT-TS to Reduce Suicide Risk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Aileen Aldalur, Assistant Professor of Psychiatry, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1K23MH137406-01A1 (NIH); 1K23MH137406-01A1 (NIH)
Record Dates: First submitted 2025-12-08; First posted 2025-12-12 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Depression - Major Depressive Disorder; Anxiety; PTSD - Post Traumatic Stress Disorder; Insomnia; Alcohol Use Disorder (AUD); Suicide Ideation
Keywords: Deaf; Mental Health; Treatment-Seeking; Suicide; Cognitive Behavioral Therapy for Treatment-Seeking
MeSH Terms: conditions — Anxiety Disorders; Combat Disorders; Sleep Initiation and Maintenance Disorders; Alcoholism; Psychological Well-Being; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist Control Group (No Intervention): During study assessments, subjects will receive a suicide risk assessment, with actions commensurate with risk level, and a list of Deaf crisis intervention resources with instructions provided on how to use them. The list of resources contains crisis hotlines that are accessible for Deaf individuals including text-based options (e.g., Crisis Text line, 988 text number) and options to talk with counselors in ASL (e.g., 988 ASL services, DeafLEAd Crisis Line). The study coordinator will review each resource and explain their use. Subjects will be emailed this list of resources after their assessment. Other brief interventions that could be provided based on subject presentation include encouraging subjects to seek social support and share their thoughts with others; elicitation of coping strategies; and lethal means safety planning.
- Deaf CBT-TS Intervention Group (Experimental): Intervention Group
  Interventions: Behavioral: Deaf CBT-TS

INTERVENTIONS:
Behavioral: Deaf CBT-TS — Deaf CBT-TS is a two-session (90 minutes each) Zoom-based intervention designed to target a change in the beliefs that influence whether or not someone initiates mental health treatment. The intervention works by modifying problematic beliefs, providing accurate information about treatment, and problem-solving barriers. The first session is structured in four phases: (1) history of symptoms and current functioning, (2) coping strategies, (3) evaluation and modification of treatment beliefs using CBT strategies, and (4) action planning. Subjects are provided a list of resources for seeking treatment, as well as a personalized search of treatment options (conducted by the interventionist) in their area based on their insurance and language preference. The second session occurs within 3 weeks and is designed to check in with subjects regarding progress on their action plan, provide assistance in identifying treatment options, and problem-solve barriers
  Arms: Deaf CBT-TS Intervention Group

SUMMARY:
The goal of this clinical trial is to learn if a short, Zoom-based intervention, Cognitive Behavioral Therapy for Treatment-Seeking for Deaf Individuals (Deaf CBT-TS) can change beliefs about mental health treatment and increase treatment-seeking behaviors in Deaf adults with untreated mental health or alcohol use problems. It will also see if Deaf CBT-TS may reduce suicide risk and explore factors that may increase the effectiveness of Deaf CBT-TS. The main questions it aims to answer are:

* Does Deaf CBT-TS increase positive beliefs about treatment and increase treatment-seeking behaviors?
* Does Deaf CBT-TS increase hope and reduce mental health symptoms, suicide ideation, and alcohol use?
* Is Deaf CBT-TS more effective for individuals with less cultural stress compared to those with high levels of cultural stress?
* Is Deaf CBT-TS more effective for Deaf individuals in residential areas with more Deaf resources than those with less Deaf resources? Researchers will compare individuals who complete Deaf CBT-TS to those on a waitlist to see if Deaf CBT-TS works to increase positive beliefs about treatment and treatment-seeking behaviors.

Participants will:

* Complete a baseline assessment including demographic information, measures of hope, general mental health and functioning, alcohol use, suicide ideation, cultural stress, and beliefs about treatment.
* Receive Deaf CBT-TS (2 sessions) or be placed on a waitlist with the option of receiving Deaf CBT-Ts after 4 months
* Complete two follow-up assessments in 2 and 4 months.

DETAILED DESCRIPTION:
The proposed project is a two-arm randomized controlled trial of a zoom-based intervention, Cognitive Behavioral Therapy for Treatment-Seeking for Deaf Individuals (Deaf CBT-TS) vs. a waitlist control, with follow-up at 2 and 4 months to assess the intervention's ability to modify beliefs about treatment (intervention principles) and increase treatment-seeking behaviors (target mechanism), as well as explore its potential to increase hope and reduce indicators of suicide risk. The investigators will also examine factors that may impact the efficacy of the intervention including levels of Deaf acculturative stress and subject residential location (Rochester, access to URMC resources vs. other locations across the U.S. with less Deaf resources). Subjects are 110 Deaf adults who report American Sign Language as their primary method of communication, have clinically significant symptoms of a mental health disorder (depression, anxiety, PTSD, insomnia, or alcohol use disorder), and are not engaged in professional mental health or alcohol specialty treatment (e.g., counseling, psychiatric services). The investigators will oversample subjects with recent suicide ideation (50%). Half of the subjects will be recruited from Rochester and the other half nationally. The Specific Aims include (1) to test whether Deaf CBT-TS engages the intervention principles and target mechanism (co-primary outcomes: changes in behavioral, normative, and control beliefs about treatment; and initiation of professional treatment); (2) to explore changes in hope and reductions in indicators of suicide risk (mental health symptoms, alcohol use, and severity of suicide ideation); and (3) to identify factors that could impact the efficacy of Deaf CBT-TS (Deaf acculturative stress and residential location).

Subjects will complete a baseline assessment including demographic information, measures of Deaf acculturative stress, hope, general mental health and functioning, alcohol use, suicide ideation, and beliefs about treatment. Subjects who complete the baseline assessment will be randomized to Deaf CBT-TS or a waitlist control, using stratified randomization based on sex assigned at birth, prior suicide attempt, and residential location (Rochester vs. other U.S. locations). During study assessments, all subjects will receive suicide risk assessments using the Columbia-Suicide Severity Rating Scale (C-SSRS), with actions commensurate with risk level, and a list of Deaf crisis intervention resources. The study coordinator will review each resource on the list and explain how to use them. Study conditions are Deaf CBT-TS (2 sessions) and waitlist control. Deaf CBT-TS involves 2 intervention sessions lasting up to 90 minutes each. The follow-up assessments (2 and 4 months) include the baseline measures of hope, general mental health and functioning, alcohol use, suicide ideation, and beliefs about treatment, as well as a treatment utilization survey to assess the subjects' use of professional mental health and alcohol specialty treatment since their last study visit. Subjects in the waitlist control group who have not engaged in professional mental health or alcohol treatment will be offered the Deaf CBT-TS intervention after their 4-month follow-up assessment.

ELIGIBILITY:
Inclusion criteria:

* adult (aged 18 years or older)
* Self-identify as Deaf or hard of hearing (any degree of hearing loss)
* Primary method of communication is American Sign Language
* Positive screen for one or more mental health disorders including depression (PHQ-9 > 10), anxiety (GAD-7 > 10), posttraumatic stress disorder (PCL-5 > 31), insomnia (ISI > 15), or alcohol use disorder (AUDIT > 16)
* No current professional mental health or alcohol specialty treatment (e.g., counseling, psychiatric services) per standardized self-report
* Access to video chat technology with internet and webcam.

Exclusion criteria:

* unable to communicate with the researcher in American Sign Language
* current alcohol withdrawal necessitating medical evaluation
* current psychiatric impairment necessitating emergency services or inpatient admission (i.e., imminent danger of harm to self or others)
* unable to comprehend the nature of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Beliefs About Treatment | Baseline to 2-month follow-up
  The Perceptions About Services Scale for the Deaf (PASS-D) will be used to assess participants' behavioral, normative, and control beliefs about treatment. The Behavioral Belief subscale has 10 items assessing advantages vs. disadvantages of seeking treatment, the Normative Belief subscale has 7 items assessing community support vs. opposition to seeking treatment, and the Control Beliefs subscale has 26 items assessing facilitators vs. barriers to seeking treatment. Each item is rated on a Likert scale ranging from 1 (Strongly Disagree) to 7 (Strongly Agree) with higher scores indicating more positive beliefs. Items for each subscale will be totaled.
Beliefs About Treatment (4 months) | Baseline to 4-month follow-up
  The Perceptions About Services Scale for the Deaf (PASS-D) will be used to assess participants' behavioral, normative, and control beliefs about treatment. The Behavioral Belief subscale has 10 items assessing advantages vs. disadvantages of seeking treatment, the Normative Belief subscale has 7 items assessing community support vs. opposition to seeking treatment, and the Control Beliefs subscale has 26 items assessing facilitators vs. barriers to seeking treatment. Each item is rated on a Likert scale ranging from 1 (Strongly Disagree) to 7 (Strongly Agree) with higher scores indicating more positive beliefs. Items for each subscale will be totaled.
Treatment Initiation | Baseline to 2-month follow-up
  A Treatment Utilization Survey will assess use of 12 treatment services, number of sessions attended, current treatment status (active vs. completed), reasons for seeking/not seeking treatment, and any barriers experienced. Treatment Initiation will be measured with a binary variable. Subjects who have attended or scheduled professional treatment services will be coded as 1 (initiated treatment) and those who have not attended or scheduled professional treatment services will be coded as 0 (not initiated).
Treatment Initiation (4 months) | Baseline to 4-month follow-up
  A Treatment Utilization Survey will assess use of 12 treatment services, number of sessions attended, current treatment status (active vs. completed), reasons for seeking/not seeking treatment, and any barriers experienced. Treatment Initiation will be measured with a binary variable. Subjects who have attended or scheduled professional treatment services will be coded as 1 (initiated treatment) and those who have not attended or scheduled professional treatment services will be coded as 0 (not initiated).

SECONDARY OUTCOMES:
Hope | Baseline to 2-months follow-up
  Hope will be assessed via the Beck Hopelessness Scale. The scale has 20 items scored as True or False. Scores of 1 or 0 are assigned to each item depending on the subject's response and the directionality of the item. The scores are summed with for a total score ranging from 0 - 20 and higher scores indicating more hopelessness.
Hope (4-months) | Baseline to 4-months follow-up
  Hope will be assessed via the Beck Hopelessness Scale. The scale has 20 items scored as True or False. Scores of 1 or 0 are assigned to each item depending on the subject's response and the directionality of the item. The scores are summed with for a total score ranging from 0 - 20 and higher scores indicating more hopelessness.
General Mental Health | Baseline to 2-months follow-up
  General mental health will be assessed via the PROMIS-29 V2.0. The scale has 29 items divided across 8 subscales. Three of the subscales are focused on general mental health: Anxiety, Depression, and Ability to Participate in Social Roles. These subscales each have four items rated on a Likert scale ranging from 1 (not at all) to 5 (very much) with higher scores indicating worse mental health functioning. Scores for each of the subscales will be summed and converted to T-scores. The T-scores for the three subscales will then be summed for a total score representing general mental health functioning.
General Mental Health (4 months) | Baseline to 4-month follow-up
  General mental health will be assessed via the PROMIS-29 V2.0. The scale has 29 items divided across 8 subscales. Three of the subscales are focused on general mental health: Anxiety, Depression, and Ability to Participate in Social Roles. These subscales each have four items rated on a Likert scale ranging from 1 (not at all) to 5 (very much) with higher scores indicating worse mental health functioning. Scores for each of the subscales will be summed and converted to T-scores. The T-scores for the three subscales will then be summed for a total score representing general mental health functioning.
Physical Functioning | Baseline to 2-month follow-up
  Physical functioning will be assessed via the PROMIS-29 V2.0. The scale has 29 items divided across 8 subscales. Five of the subscales are focused on physical functioning: Physical Function, Fatigue, Sleep Disturbance, Pain Interference, and Pain Intensity. The subscales Physical Function, Fatigue, Sleep Disturbance, Pain Interference each have four items rated on a Likert scale ranging from 1 (not at all) to 5 (very much) with higher scores indicating worse physical functioning. The Pain Interference subscale is a single item rated on a Likert scale ranging from 0 (no pain) to 10 (worst imaginable pain). Scores for each of the subscales will be summed and converted to T-scores. The T-scores for the five subscales will then be summed for a total score representing physical functioning.
Physical Functioning (4 months) | Baseline to 4-month follow-up
  Physical functioning will be assessed via the PROMIS-29 V2.0. The scale has 29 items divided across 8 subscales. Five of the subscales are focused on physical functioning: Physical Function, Fatigue, Sleep Disturbance, Pain Interference, and Pain Intensity. The subscales Physical Function, Fatigue, Sleep Disturbance, Pain Interference each have four items rated on a Likert scale ranging from 1 (not at all) to 5 (very much) with higher scores indicating worse physical functioning. The Pain Interference subscale is a single item rated on a Likert scale ranging from 0 (no pain) to 10 (worst imaginable pain). Scores for each of the subscales will be summed and converted to T-scores. The T-scores for the five subscales will then be summed for a total score representing physical functioning.
Alcohol Use | Baseline to 2-month follow-up
  The National Survey on Drug Use and Health (NSDUH) 30-day alcohol consumption will be used to assess alcohol use including total number of drinking days, number of drinks per drinking day, and number of heavy episodes of drinking.
Alcohol Use (4 months) | Baseline to 4-month follow-up
  The National Survey on Drug Use and Health (NSDUH) 30-day alcohol consumption will be used to assess alcohol use including total number of drinking days, number of drinks per drinking day, and number of heavy episodes of drinking.
Suicide Ideation | Baseline to 2-month follow-up
  Suicide Ideation will be assessed via the Depressive Symptom Index Suicidality Scale. The scale has four items rated on a Likert scale from 0 - 3, with higher scores indicating a higher intensity of suicide ideation.
Suicide Ideation (4 months) | Baseline to 4-month follow-up
  Suicide Ideation will be assessed via the Depressive Symptom Index Suicidality Scale. The scale has four items rated on a Likert scale from 0 - 3, with higher scores indicating a higher intensity of suicide ideation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No